CLINICAL TRIAL: NCT00680043
Title: AFX01-15: A Phase 2, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Peginesatide for the Correction of Anemia in Patients With Chronic Renal Failure (CRF) Undergoing Hemodialysis and Not on Erythropoiesis Stimulating Agent (ESA) Treatment
Brief Title: Safety & Efficacy of Peginesatide for Treatment of Anemia in Participants on Dialysis Not Receiving an ESA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affymax (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-15
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Anemia; Chronic Renal Failure; Chronic Kidney Disease
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — peginesatide; hematide; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Peginesatide 0.04 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Peginesatide 0.08 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Epoetin Alfa (Active Comparator)
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: peginesatide — Participants received peginesatide by intravenous injection once every 4 weeks at the starting dose of 0.04 milligram per kilogram (mg/kg); the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.04 mg/kg
Drug: peginesatide — Participants received peginesatide by intravenous injection once every 4 weeks at the starting dose of 0.08 mg/kg; the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.08 mg/kg
Drug: Epoetin Alfa — Participants received Epoetin alfa by intravenous injection three times a week at the starting dose of 50 Units/kg. The dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Eprex
  Arms: Epoetin Alfa

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of peginesatide for the treatment of anemia in participants with chronic kidney disease who are on dialysis and are not taking any treatment to increase their red blood cell production.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents (ESAs) have been established as a treatment for anemia in chronic renal failure subjects, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia in patients with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Eligible participants were randomized in equal proportions to two peginesatide treatment regimens, in which participants received peginesatide once every 4 weeks, and one control, epoetin alfa, treatment regimen, in which participants received epoetin alfa three times per week. Total commitment time of this study was a 4 week screening period followed by a minimum of 7 months of treatment.

ELIGIBILITY:
Inclusion Criteria

1. On hemodialysis for chronic renal failure for at least 2 weeks prior to randomization.
2. Two consecutive hemoglobin values of ≥ 8.0 g/dL and < 11.0 g/dL within the 4 weeks prior to randomization.

Exclusion Criteria

1. Females who are pregnant or breast-feeding.
2. Prior treatment with an erythropoiesis stimulating agent (ESA) in the 12 weeks prior to randomization.
3. Known intolerance to any ESA, parenteral iron supplementation, or pegylated molecule.
4. Known bleeding or coagulation disorder.
5. Known hematologic disease or cause for anemia other than renal disease
6. Poorly controlled hypertension.
7. Evidence of active malignancy within one year.
8. A scheduled kidney transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (11):
- Russia (11):
  - Research Facility, Irkutsk
  - Research Facility, Krasnodar
  - Research Facility, Krasnoyarsk
  - Research Facility, Moscow
  - Research Facility, Nizhny Novgorod
  - Research Facility, Omsk
  - Research Facility, Petrozavodsk
  - Research Facility, Saint Petersburg
  - Research Facility, Saratov
  - Research Facility, Tver'
  - Research Facility, Volzhsk

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginesatide 0.04 mg/kg: Participants received peginesatide by intravenous injection once every 4 weeks at the starting dose of 0.04 milligram per kilogram (mg/kg); the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
- Peginesatide 0.08 mg/kg: Participants received peginesatide by intravenous injection once every 4 weeks at the starting dose of 0.08 mg/kg; the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
- Epoetin Alfa: Participants received Epoetin alfa by intravenous injection three times a week at the starting dose of 50 Units/kg; the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
Period: Overall Study
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa
Started | 39 | 37 | 38
Completed | 37 | 36 | 34
Not Completed | 2 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Patient Not Compliant With Study Reqs. | 0 | 1 | 0
Not completed — Renal Transplant | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa | Total
Number analyzed (Participants) | 39 | 37 | 38 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 31 | 30 | 98
  >=65 years | 2 | 6 | 8 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.71) | 48.8 (13.55) | 51.4 (14.16) | 49.7 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 19 | 45
  Male | 27 | 23 | 19 | 69

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The baseline hemoglobin value is defined as the mean of the two most recent hemoglobin values taken prior to the day of randomization plus the value obtained on the day of randomization prior to Dose 1. The mean hemoglobin during the Evaluation period for each participant is calculated as the mean of the available hemoglobin values during Study Weeks 21 through 28.
Time Frame: Baseline and Weeks 21-28
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa
Number analyzed (Participants) | 39 | 37 | 38
g/dL
  Baseline [N=39, 37, 38] | 9.34 (0.738) | 9.20 (0.701) | 9.07 (0.739)
  Evaluation Period [N=37, 37, 36] | 11.45 (1.101) | 11.59 (0.943) | 11.49 (0.775)
  Change from Baseline [N=37, 37, 36] | 2.15 (1.038) | 2.39 (0.974) | 2.41 (0.991)
Statistical Analysis 1: Comparison: Peginesatide 0.04 mg/kg vs Epoetin Alfa; Test type: Superiority or Other; ANOVA; Least Squares Mean Difference = -0.25, 97.5% CI 2-sided [-0.79 to 0.29], Standard Error of Mean 0.238
Statistical Analysis 2: Comparison: Peginesatide 0.08 mg/kg vs Epoetin Alfa; Test type: Superiority or Other; ANOVA; Least Squares Mean Difference = -0.02, 97.5% CI 2-sided [-0.56 to 0.52], Standard Error of Mean 0.238

2. Secondary Outcome: Proportion of Participants Who Receive Red Blood Cell (RBC) or Whole Blood Transfusions During the Correction and Evaluation Periods
Time Frame: Weeks 1 to 28
Population: Full Analysis Population
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa
Number analyzed (Participants) | 39 | 37 | 38
percentage of participants | 0.026 | 0.0 | 0.0

3. Secondary Outcome: Proportion of Participants Achieving Hemoglobin Response During the Correction and Evaluation Periods
Description: A hemoglobin response is defined as a hemoglobin increase of ≥ 1.0 g/dL above baseline and a hemoglobin ≥ 11.0 g/dL without RBC or whole blood transfusion during the previous 8 weeks.
Time Frame: Weeks 1 to 28
Population: Full Analysis Population
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa
Number analyzed (Participants) | 39 | 37 | 38
percentage of participants | 0.923 | 0.973 | 1.0
Statistical Analysis 1: Comparison: Peginesatide 0.04 mg/kg vs Epoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.84 to 1.01]
Statistical Analysis 2: Comparison: Peginesatide 0.08 mg/kg vs Epoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.92 to 1.03]

ADVERSE EVENTS:
Arm/Group | Peginesatide 0.04 mg/kg | Peginesatide 0.08 mg/kg | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 6/39 | 8/37 | 4/38
Other Adverse Events (participants affected / at risk) | 21/39 | 26/37 | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.04 mg/kg (N=39) | Peginesatide 0.08 mg/kg (N=37) | Epoetin Alfa (N=38)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic vascular disorder (Vascular disorders) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.04 mg/kg (N=39) | Peginesatide 0.08 mg/kg (N=37) | Epoetin Alfa (N=38)
Angina pectoris (Cardiac disorders) | 1 | 1 | 4
Palpitations (Cardiac disorders) | 1 | 0 | 2
Hyperparathyroidism secondary (Endocrine disorders) | 3 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Catheter site inflammation (General disorders) | 1 | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 3 | 3 | 1
Influenza (Infections and infestations) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 5
Procedural hypotension (Injury, poisoning and procedural complications) | 9 | 4 | 8
Procedural hypertension (Injury, poisoning and procedural complications) | 5 | 4 | 6
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0
Blood pressure increased (Investigations) | 1 | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 2
Transaminases increased (Investigations) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 7 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 3 | 3 | 5
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 1 | 5
Hypertension (Vascular disorders) | 9 | 6 | 5
Hypotension (Vascular disorders) | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the primary safety and efficacy results will include data from all appropriate study sites. Either after the first multicenter publication, or following 36 months after the completion of the study, Investigators are free to publish; such publications may not contain Sponsor Confidential Information and may be subject to Sponsor review 60 days prior to submission for publication.